CLINICAL TRIAL: NCT00673478
Title: A Randomised, Open-label, 4-way Crossover Study to Characterize the Pharmacokinetics, Safety and Efficacy of FDC Tiotropium/Salmeterol, Tiotropium, Salmeterol and a Free Combination of Tiotropium Plus Salmeterol Following 4-week Treatment Periods in Patients With COPD.
Brief Title: Tiotropium and Salmeterol PK Study in COPD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Crossover | Purpose: Treatment
Other Study IDs: 1184.24; EudraCT 2007-000207-15
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Salmeterol Xinafoate; Tiotropium Bromide

INTERVENTIONS:
Drug: Tiotropium+Salmeterol
Drug: Salmeterol
Drug: Tiotropium

SUMMARY:
The primary objective of this study is to characterize the pharmacokinetics (i.e. systemic exposure to tiotropium and salmeterol) of tiotropium qd + salmeterol qd or bid versus tiotropium qd and salmeterol bid following 4-week treatment periods in patients with chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

COPD patients of >= 40 years old with moderate to severe COPD who are current or ex-smokers with a smoking history of at least 10 pack-years

Exclusion Criteria:

1. Recent history of myocardial infarction, life-threatening cardiac arrhythmia or hospitalisation for cardiac failure
2. History of asthma
3. Malignancy requiring treatment within past 5 years
4. Life-threatening pulmonary obstruction, cystic fibrosis or clinically evident bronchiectasis
5. Known active tuberculosis
6. Pregnant or nusing women
7. Known hypersensitivity to components of the study medication

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC0-∞ ) of tiotropium in plasma | 16 weeks
Maximum measured concentration of tiotropium in plasma (Cmax) | 16 weeks
Amount of tiotropium that was eliminated in urine (Ae0-8) from time point 0 to 8 hours post-inhalation | 16 weeks
AUC0-∞ of salmeterol in plasma | 16 weeks
Cmax salmeterol in plasma | 16 weeks

SECONDARY OUTCOMES:
Area under the concentration time curve (AUCt1-t2) of tiotropium and salmeterol in plasma over the time interval t1 to t2 for time intervals 0 to 4, 0 to 6, and 0 to 8 hours after inhalation (AUC0-4, AUC0-6, and AUC0-8) | 16 weeks
Time from dosing to the maximum concentration of tiotropium and salmeterol in plasma (tmax) | 16 weeks
Terminal rate constant in plasma (λz) | 16 weeks
Terminal half-life (t½) of tiotropium and salmeterol in plasma) | 16 weeks
Mean residence time (MRTih) of tiotropium and salmeterol in the body after inhalational administration | 16 weeks
Apparent clearance (CL/F) of tiotropium and salmeterol in plasma after extravascular administration) | 16 weeks
Apparent volume of distribution (Vz/F) during the terminal phase (λz) following an extravascular dose) | 16 weeks
Amount of tiotropium that is eliminated in urine from the time point t1 to time point t2 (Aet1-t2) (Ae0-2, Ae2-4, Ae4-8, Ae0-8) | 16 weeks
Fraction of tiotropium eliminated in urine from time point t1 to time point t2 (fet1-t2) (fe0-2, fe2-4, fe4-8, fe0-8) | 16 weeks
Renal clearance of tiotropium from the time point t1 until the time point t2 (CLR,t1-t2) (CLR,0-2, CLR, 2-4, CLR,4-8, CLR,0-8) | 16 weeks
All adverse events | 20 weeks
Blood pressure (seated) recorded in conjunction with 12-lead ECG recordings pre-dose and following the morning dose of randomized treatment | 20 weeks
Number of patients with abnormalities in routine blood chemistry, haematology and urinalysis | 16 weeks
Trough forced expiratory volume in one second (FEV1) | 16 weeks
Trough forced vital capacity (FVC) | 16 weeks
FEV1 area under the curve 0 to 8 hours (FEV1 AUC0-8h) | 16 weeks
FVC area under the curve 0 to 8 hours (FVC AUC0-8h) | 16 weeks
Individual FEV1and FVC measurements at each time point at the end of each 4-week treatment period. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- Belgium (2):
  - 1184.24.32001 Boehringer Ingelheim Investigational Site, Genk
  - 1184.24.32002 Boehringer Ingelheim Investigational Site, Hasselt
- 1184.24.31001 Boehringer Ingelheim Investigational Site, Heerlen, Netherlands

REFERENCES:
- [Derived] Parigi TL, Nardone OM, Lisa M, Massimino L, Gabbiadini R, Innocenti T, Bertani L, Del Gaudio A, Florez P, Bertin L, Barberio B, Hupe M, Lopetuso L, Allocca M, D'Amico F, Furfaro F, Zilli A, Fiorino G, Ungaro F, Castiglione F, Savarino E, Dragoni G, Scaldaferri F, Armuzzi A, Peyrin-Biroulet L, Jairath V, Pizarro TT, Danese S. The Impact of E-Cigarettes and Heat-Not-Burn Tobacco on Postoperative Recurrence of Crohn's Disease: A Multicenter International Study. Am J Gastroenterol. 2025 Oct 24. doi: 10.14309/ajg.0000000000003810. Online ahead of print. PMID 41134080